CLINICAL TRIAL: NCT00644943
Title: A Comparison of the Safety and Efficacy of Cefdinir Oral Suspension Versus Amoxicillin/Clavulanate in Pediatric Subjects With Acute Otitis Media
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Angela M Nilius, Ph.D., Abbott
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: M02-541
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Cefdinir; Amoxicillin

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: cefdinir (Omnicef)
- 2 (Active Comparator)
  Interventions: Drug: amoxicillin

INTERVENTIONS:
Drug: cefdinir (Omnicef) — oral suspension (7 mg/kg, ql2hr) for 5 days
  Other Names: ABT-198; Omnicef; cefdinir
  Arms: 1
Drug: amoxicillin — oral suspension (45 mg/kg/day, q l2 hours) for 10 days
  Arms: 2

SUMMARY:
The primary objective is to compare the safety and efficacy of cefdinir oral suspension, 7 mg/kg/day ql2hrs for 5 days, to amoxicillin/clavulanate oral suspension 45 mg/kg/day (based on amoxicillin component), in divided doses, q12h for 10 days, in children between 6 months and 6 years of age, with AOM.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis, documented by medical history and physical examination, is acute otitis media <=1 week
* Clinical signs and symptoms include >=1 of the following: ear pain; ear fullness, decreased hearing, or discharge from the external auditory canal (following acute perforation of the tympanic membrane).
* At least two of the following conditions are present in at least one ear: bulging tympanic membrane, which may have redness; loss of the normal light reflex and tympanic membrane landmarks and abnormal tympanic membrane mobility on biphasic pneumatic otoscopy, due to the presence of pus or fluid behind it and edema of the tympanic membrane.
* Have evidence of middle ear fluid demonstrated by acoustic reflect-tympometry.
* Generally in good health based on medical history, vital signs, physical exam, and historical laboratory results

Exclusion Criteria:

* Previous enrollment in this study.
* Enrollment in any other investigational study using unapproved products or unapproved doses, including investigational vaccines in the previous four weeks prior to study start.
* Hypersensitivity reactions to cefdinir, other cephalosporins, penicillins, other drugs, and/or sensitivity to multiple allergens.
* Presence of tympanostomy tubes or otitis externa at Evaluation 1.
* Systemic treatment with any anti-infective agent within 7 days (14 days for azithromycin) prior to Evaluation 1 or during the study.
* Treatment with a long-acting injectable antimicrobial agent (e.g., penicillin G benzathine) within 4 weeks prior to study drug administration.
* Concomitant infection, that requires additional antimicrobial therapy.
* Evidence of chronic, suppurative otitis media.
* Evidence of a physiologic, anatomic, or immunologic defect, which would interfere with resolution of this episode of acute otitis media.
* Presence of a disease, complicating factor (e.g., mastoiditis), or structural abnormality that would preclude evaluation of the subject's therapeutic response.
* Known, severe renal impairment (i.e., creatinine clearance < 30 mUmid1.73 m2).
* History of Augmentin-associated cholestatic jaundicehepatic dysfunction.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 425 (Actual)
Dates: Start 2003-02; Primary Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Clinical Cure Rate | 9 days

SECONDARY OUTCOMES:
Sustained Clinical Cure Rate | 28 days

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Ozark, Alabama
  - Mesa, Arizona
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Clovis, California
  - Fresno, California
  - Longmont, Colorado
  - Fairfield, Connecticut
  - Marietta, Georgia
  - Stone Mountain, Georgia
  - Bardstown, Kentucky
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Ruston, Louisiana
  - Shreveport, Louisiana
  - Kalamazoo, Michigan
  - Richland, Michigan
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Columbus, Ohio
  - Medford, Oregon
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Lake Jackson, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Vienna, Virginia